CLINICAL TRIAL: NCT02625181
Title: Real-time Decision Support for Postoperative Nausea and Vomiting (PONV) Prophylaxis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Jonathan Wanderer, Medical Director of Procedure Preparation Center, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 151750
Record Dates: First submitted 2015-11-12; First posted 2015-12-09 (Estimated); Results first posted 2019-03-07 (Actual); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Postoperative Nausea and Vomiting
Keywords: Decision support; Prediction models; PONV; prophylaxis; Decision Support Systems, Clinical; Decision Support Techniques
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Anesthesia, General; Elective Surgical Procedures; Propofol; Sevoflurane; Isoflurane; Desflurane; Scopolamine; Droperidol; Haloperidol; Dexamethasone; Promethazine; Meclizine; Aprepitant; Metoclopramide; Fentanyl; Sufentanil; Alfentanil; Remifentanil; Morphine; Meperidine; Hydromorphone; Methadone; Oxycodone; Oxymorphone; Hydrocodone; Ketamine; Ondansetron; Granisetron; dolasetron; Palonosetron; Tropisetron; ramosetron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- PONV clinical decision support system (Experimental): Automated recommendations on PONV prophylaxis provided to anesthesia providers through the anesthesia information management system and email.
  Interventions: Procedure: Automated recommendation at the start of the case; Procedure: Automated notification at the start of surgery; Procedure: Preoperative recommendations: by email; Procedure: Automated notification at the end of surgery; Device: Anesthesia Information Management System (AIMS); Device: Perioperative Data Warehouse (PDW); Procedure: General anesthesia; Procedure: Elective surgery; Drug: Propofol; Drug: Sevoflurane; Drug: Isoflurane; Drug: Desflurane; Drug: Scopolamine; Drug: Droperidol; Drug: Haloperidol; Drug: Dexamethasone; Drug: Promethazine; Drug: Meclizine; Drug: Aprepitant; Drug: Metoclopramide; Drug: Fentanyl; Drug: Sufentanil; Drug: Alfentanil; Drug: Remifentanil; Drug: Morphine; Drug: Meperidine; Drug: Hydromorphone; Drug: Methadone; Drug: Oxycodone; Drug: Oxymorphone; Drug: Hydrocodone; Drug: Ketamine; Drug: Ondansetron; Drug: Granisetron; Drug: Dolasetron mesylate; Drug: Palonosetron; Drug: Tropisetron; Drug: Ramosetron

INTERVENTIONS:
Procedure: Automated recommendation at the start of the case — The first notification is the main notification that informs the anesthesia providers at the start of anesthesia of the risk score for that individual patient and the recommended number of prophylactic interventions. The notification occurs within the anesthesia information management system (AIMS)
Procedure: Automated notification at the start of surgery — The second notification within the AIMS will notify the anesthesia providers at the start of surgery when no prophylaxis has been given while three or more interventions were recommended.
Procedure: Preoperative recommendations: by email — A recommendation on PONV prophylaxis to anesthesia providers through email at the Vanderbilt University Medical Center.
Procedure: Automated notification at the end of surgery — A notification will remind anesthesia providers at the closing of surgery how many prophylactic interventions are required to adhere to the recommended number of interventions.
Device: Anesthesia Information Management System (AIMS) — The anesthesia electronic record keeping system
Device: Perioperative Data Warehouse (PDW) — The data warehouse that is used to gather perioperative data and create user reports. In this instance the PDW will be used to send the preoperative emails.
Procedure: General anesthesia — Any anesthetic drugs that are used to induce general anesthesia above the level of sedation.
Procedure: Elective surgery — Surgical procedures that are scheduled and not an emergency.
Drug: Propofol — Anesthetic drug used to maintain general anesthesia
Drug: Sevoflurane — Anesthetic drug used to maintain general anesthesia
Drug: Isoflurane — Anesthetic drug used to maintain general anesthesia
Drug: Desflurane — Anesthetic drug used to maintain general anesthesia
Drug: Scopolamine — Prophylactic antiemetic
Drug: Droperidol — Prophylactic antiemetic & rescue antiemetic
Drug: Haloperidol — Prophylactic antiemetic & rescue antiemetic
Drug: Dexamethasone — Prophylactic antiemetic & rescue antiemetic
Drug: Promethazine — Prophylactic antiemetic & rescue antiemetic
Drug: Meclizine — Prophylactic antiemetic & rescue antiemetic
Drug: Aprepitant — Prophylactic antiemetic & rescue antiemetic
Drug: Metoclopramide — Rescue antiemetic
Drug: Fentanyl — Analgesic drug / Opioid
Drug: Sufentanil — Analgesic drug / Opioid
Drug: Alfentanil — Analgesic drug / Opioid
Drug: Remifentanil — Analgesic drug / Opioid
Drug: Morphine — Analgesic drug / Opioid
Drug: Meperidine — Analgesic drug / Opioid
Drug: Hydromorphone — Analgesic drug / Opioid
Drug: Methadone — Analgesic drug / Opioid
Drug: Oxycodone — Analgesic drug / Opioid
Drug: Oxymorphone — Analgesic drug / Opioid
Drug: Hydrocodone — Analgesic drug / Opioid
Drug: Ketamine — Analgetic / Analgesic drug
Drug: Ondansetron — Prophylactic antiemetic & rescue antiemetic
Drug: Granisetron — Prophylactic antiemetic & rescue antiemetic
Drug: Dolasetron mesylate — Prophylactic antiemetic & rescue antiemetic
Drug: Palonosetron — Prophylactic antiemetic & rescue antiemetic
Drug: Tropisetron — Prophylactic antiemetic & rescue antiemetic
Drug: Ramosetron — Prophylactic antiemetic & rescue antiemetic

SUMMARY:
The purpose of this study is to determine how automated recommendations are best presented to optimize the adherence to guidelines on prophylaxis for nausea and vomiting after surgery.

DETAILED DESCRIPTION:
Nausea and vomiting after surgery (PONV) is a common side effect of the surgical procedure, general anesthesia and opioid use occurring in about one third of patients. In addition to being very unpleasant for patients, it is associated with longer recovery room stays and increased costs. Much research has been done on prophylactic interventions that may be applied during the surgical procedure to prevent PONV. Current national guidelines recommend that a risk score is used to decide on the number of prophylactic interventions to administer to a patient. Based on specific characteristics of individual patients and the procedures that they are about to undergo, such a risk score predicts the risk of PONV for each individual. According to the national guidelines, patients with higher risks of PONV should receive more prophylactic interventions. However, in a busy operating room where the anesthesia provider performs multiple patient care tasks, closely following the recommendations to minimize the risk of PONV is often difficult.

Computers may help anesthesia providers to adhere to best practices for PONV prevention by providing so-called decision support. A decision support system for PONV automatically calculates the risk of PONV for an individual patient and presents this predicted risk to the anesthesia provider on the computer screen that is being used by the anesthesia team for record keeping. In recent studies, such decision support systems have been demonstrated to improve adherence to PONV guidelines, especially when a recommendation on the number of interventions is added to the predicted risk. However, in these studies there was still quite some room for improvement of the adherence to PONV guidelines. In general, implementation science is only beginning to understand how such decision support systems are best used to improve medical decision making and minimize practice variations among providers. Further study of how the design of decision support systems impacts the decision making of healthcare providers is therefore warranted.

In this proposed study, the investigators will implement several decision support elements for PONV that aim to help anesthesia providers to adhere to the departmental PONV guidelines during the anesthetic case. The study consists of three phases. The first phase is the preintervention phase - i.e. before the decision support has been implemented. The second phase is the first intervention phase with one CDSS feature added. The third phase is the second intervention phase with another CDSS feature added.

The decision support elements will provide information about the patient's predicted risk of PONV and the number of prophylactic interventions that the departmental guidelines recommend based on that risk. We will start with preoperative email notifications, followed by an element within the anesthesia information management system (AIMS) that are displayed around the start and end of the procedure. All forms of decision support only provide recommendations. The anesthesia provider is free to act on the message or ignore the notifications.

The investigators will compare the adherence to PONV guidelines and the actual occurrence of PONV (both nausea and emetic events: vomiting and retching) in the post-anesthesia care unit (PACU) between all study phases and between the different interventions. The goal of the comparison is to evaluate which decision support elements have an added value to optimize guideline adherence for PONV prophylaxis.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients (18 years and older) that are scheduled for an elective surgical procedure under general anesthesia

Exclusion Criteria:

* Patients undergoing emergency surgery or organ transplantation
* Patients that are transferred directly to the Intensive Care Unit after the end of the procedure
* Patients that die intraoperatively
* Procedures that only require a sedative level of anesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27034 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-11-02 (Actual); Study Completion 2017-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan P Wanderer, MD, MPhil, Principal Investigator — Vanderbilt University Medical Center, Division of Anesthesiology
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Baseline Measurement: No recommendations were provided for PONV prophylaxis.
- CDS Email Recommendations: Automated recommendations on PONV prophylaxis provided by email only.
- CDS Email + Real TIme Recommenations: Number of interventions for PONV prophylaxis were provided both by real-time clinical decision support and via email.
Period: Overall Study
Arm/Group | Baseline Measurement | CDS Email Recommendations | CDS Email + Real TIme Recommenations
Started (Baseline measurement period) | 1518 | 12809 | 12707
Completed | 1518 | 12809 | 12707
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: This population was analyzed prior to the institution of CDS for PONV prophylaxis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Baseline Measurement | CDS Email Recommendations | CDS Email + Real TIme Recommenations | Total
Number analyzed (Participants) | 1518 | 12809 | 12707 | 27034
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1131 | 9573 | 9603 | 20307
  >=65 years | 387 | 3236 | 3104 | 6727
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (16.78) | 52 (16.73) | 51 (17.15) | 52 (16.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 813 | 6550 | 6212 | 13575
  Male | 705 | 6259 | 6495 | 13459
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 12 | 23 | 38
  Asian | 11 | 100 | 110 | 221
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 170 | 1321 | 1595 | 3086
  White | 1279 | 10823 | 10498 | 22600
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 55 | 553 | 481 | 1089
Region of Enrollment [Number; unit: participants]
  United States | 1518 | 12809 | 12707 | 27034
History of PONV/Motion Sickness [Count of Participants; unit: Participants] | 226 | 2303 | 10728 | 13257
Smoking Status is Current Non Smoker [Count of Participants; unit: Participants] | 1183 | 9723 | 9352 | 20258

OUTCOME MEASURES:

1. Primary Outcome: Adherence to PONV Guidelines
Description: PONV guideline adherence: percentage of patients who received the exact number of prophylactic interventions for PONV that were recommended by the decision support.
Time Frame: A specific time frame on the day of surgery: the start of admission at the holding room to the end of the anesthetic case
Measure: Count of Participants; unit: Participants
Arm/Group | Baseline Measurement | CDS Email Recommendations | CDS Email + Real TIme Recommenations
Number analyzed (Participants) | 1518 | 12809 | 12707
Participants | 666 | 5260 | 5863

2. Secondary Outcome: PONV Incidence: Number of Participants With Postoperative Nausea and Vomiting
Description: The occurrence of PONV, as defined by the administration of antiemetics in the PACU between admission to PACU and discharge from PACU.
Time Frame: PACU recovery period
Measure: Count of Participants; unit: Participants
Arm/Group | Baseline Measurement | CDS Email Recommendations | CDS Email + Real TIme Recommenations
Number analyzed (Participants) | 1518 | 12809 | 12707
Participants | 139 | 1323 | 1343

3. Secondary Outcome: The Number of Prophylactic Interventions for PONV
Description: the absolute number of prophylactic interventions applied between the admission of the patient in the holding room until admission to the PACU.
Time Frame: A specific time frame on the day of surgery: from the start of admission at the holding room to the end of the anesthetic case
Measure: Mean (Standard Deviation); unit: prophylactic antiemetics administered
Arm/Group | Baseline Measurement | CDS Email Recommendations | CDS Email + Real TIme Recommenations
Number analyzed (Participants) | 1518 | 12809 | 12707
prophylactic antiemetics administered | 2.196 (0.932) | 2.176 (0.988) | 2.129 (0.977)

4. Secondary Outcome: Time to Discharge From the Postanesthesia Care Unit (PACU)
Description: This is the number of minutes from admission to the PACU until discharge, assessed up to 2 days
Time Frame: A specific time frame on the day of surgery: from the start of admission to the PACU to discharge from the PACU
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Baseline Measurement | CDS Email Recommendations | CDS Email + Real TIme Recommenations
Number analyzed (Participants) | 1518 | 12809 | 12707
minutes | 266 (374) | 264 (371) | 266 (361)

ADVERSE EVENTS:
Time Frame: We analyzed adverse events in this patient population during their intraoperative course from entry into OR until exit from the OR (adverse events sourced from our adverse event reporting system), and during their hospitalization (source for mortality data), an average of 4.9 days.
Description: We utilized our perioperative information management system to determine the number of adverse events that occurred associated with the patients' intraoperative course. We used our hospital registration system to determine all cause mortality for this patient population.
Groups:
- PONV Clinical Decision Support System: Automated recommendations on PONV prophylaxis provided to anesthesia providers through the anesthesia information management system and email.
  Automated recommendation at the start of the case: The first notification is the main notification that informs the anesthesia providers at the start of anesthesia of the risk score for that individual patient and the recommended number of prophylactic interventions. The notification occurs within the anesthesia information management system (AIMS)
  Preoperative recommendations: by email: A recommendation on PONV prophylaxis to anesthesia providers through email.
Arm/Group | PONV Clinical Decision Support System
All-Cause Mortality (participants affected / at risk) | 90/27034
Serious Adverse Events (participants affected / at risk) | 90/27034
Other Adverse Events (participants affected / at risk) | 0/27034
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | PONV Clinical Decision Support System (N=27034)
Mortality - Baseline (Investigations) | 7/1518 (7)
Mortality - CDS Email Recommendations (Investigations) | 43/12809 (43)
Mortality - CDS Email + Real Time Recommendations (Investigations) | 40/12707 (40)

LIMITATIONS AND CAVEATS:
We were unable to complete analysis of hyperlink data for PONV recommendations as planned because the data were not archived as intended. We were unable to include University of Washington as a collaborative site due to technical differences.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-28): https://cdn.clinicaltrials.gov/large-docs/81/NCT02625181/Prot_SAP_000.pdf